CLINICAL TRIAL: NCT02014844
Title: An Open-Label Pilot Phase 2 Study to Investigate the Preliminary Efficacy and Safety of Aldoxorubicin in Subjects With Unresectable Glioblastoma Whose Tumors Have Progressed Following Prior Treatment With Surgery, Radiation and Temozolomide
Brief Title: Phase 2 Study to Investigate the Efficacy and Safety of Aldoxorubicin in Subjects With Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALDOXORUBICIN-P2-GBM-01
Record Dates: First submitted 2013-12-09; First posted 2013-12-18 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2015-09

CONDITIONS: Glioblastoma
Keywords: glioblastoma; aldoxorubicin; temozolomide; brain cancer; brain tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — DOXO-EMCH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 250 mg/m2 aldoxorubicin (Experimental): Subjects received 250 mg/m2 aldoxorubicin IV.
  Interventions: Drug: 250 mg/m2 aldoxorubicin
- 350 mg/m2 aldoxorubicin (Experimental): Subjects received 350 mg/m2 aldoxorubicin IV.
  Interventions: Drug: 350 mg/m2 aldoxorubicin

INTERVENTIONS:
Drug: 250 mg/m2 aldoxorubicin
  Other Names: INNO-206
  Arms: 250 mg/m2 aldoxorubicin
Drug: 350 mg/m2 aldoxorubicin
  Other Names: INNO-206
  Arms: 350 mg/m2 aldoxorubicin

SUMMARY:
This is a pilot study to determine the efficacy and safety of aldoxorubicin in subjects with glioblastoma who have progressed following surgery and prior treatments.

DETAILED DESCRIPTION:
This is a second line open-labeled pilot phase 2 study in subjects with glioblastoma whose tumors have progressed following prior treatment with surgery, radiation and Temozolomide. Patients who have received avastin as a second-line treatment are not eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older; male or female
2. Histologically or cytologically confirmed unresectable GBM. Subjects with recurrent disease whose prior pathology demonstrated GBM will not need to be re-biopsied. Subjects with prior low-grade glioma or anaplastic glioma are eligible if histological assessment demonstrates transformation into GBM.
3. Cancer progression after treatment with the following: surgery, radiation therapy and temozolomide as first line treatment with no other therapy prior to tumor recurrence.

   1. Radiographic progression by RANO Working Group Criteria will be confirmed by Imaging Endpoints, a central imaging vendor.
   2. By tumor biopsy if conducted within 4 weeks of randomization.
4. An interval of at least 12 weeks after last dose of radiation and temozolomide is required, unless cancer progression is proven by diagnostic tumor biopsy. If temozolomide is being used in a maintenance phase, there must be a 28-day washout period prior to Randomization.
5. Stable or decreasing dose of corticosteroids for at least 7 days prior to randomization.
6. Capable of providing informed consent and complying with trial procedures.
7. Karnofsky Performance Status 70 or above.
8. ECOG performance status 0-2.
9. Life expectancy 8 or more weeks.
10. Measurable tumor lesions according to RANO working Group Criteria.

    a. In the case that there is "non-measurable" disease due to a radical surgical resection during screening, the subject still qualifies if Inclusion #3(b) is met.
11. Women must not be able to become pregnant for the duration of the study.
12. Women of childbearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
13. Geographically accessible to site, i.e. the ability to come to the study site for each scheduled appointment and evaluation.

Exclusion Criteria:

1. Prior exposure to the an anthracycline.
2. Any therapeutic regimen for treatment of recurrent tumor after first line treatment with surgery, radiation and temozolomide.
3. Prior treatment with bevacizumab or an experimental anti-angiogenic agent.
4. Palliative surgery and/or radiation treatment less than 4 weeks to randomization.
5. Exposure to any investigational agent within 30 days of Randomization.
6. History of other malignancies (except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix) unless documented free of cancer for 3 or more years.
7. Laboratory values: screening serum creatinine > 1.5xULN, ALT > 2.5xULN, total bilirubin > 1.5xULN, ANC < 1500/mm3, platelet concentrations < 100,000/mm3, absolute lymphocyte count < 1000/mm3, hematocrit level < 27% for females or < 30% for males, serum albumin ≤ 2.5 g/dL, PT/INR 1.5xULN or >3xULN on anticoagulant with no evidence of active bleeding.
8. Evidence of CNS hemorrhage CTCAE ≥ grade 2 on baseline MRI.
9. Clinically evident congestive heart failure > class II of the NYHA guidelines.
10. Current, serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrythmias classified as Lown III, IV or V.
11. History or signs of active coronary artery disease with or without angina pectoris.
12. Serious myocardial dysfunction defined as ultrasound-determined LVEF < 45% of predicted institutional normal value.
13. Baseline ATc>470 msec and/or previous history of QT prolongation.
14. Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals, or anti-fungals.
15. History of HIV infection.
16. Major surgery, except diagnostic tumor biopsy, within 4 weeks of randomization.
17. Any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
18. Any condition that is unstable and could jeopardize the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Ochsner Health System, New Orleans, Louisiana
  - Texas Oncology-Austin Midtown, Austin, Texas

REFERENCES:
- See also: Related Info — https://news.yahoo.com/aldoxorubicin-continues-demonstrate-positive-clinical-140059672.html?guccounter=1

RESULTS

PARTICIPANT FLOW:
Groups:
- 250 mg/m^2 Aldoxorubicin: Subjects received 250 mg/m^2 aldoxorubicin IV.
- 350 mg/m^2 Aldoxorubicin: Subjects received 350 mg/m^2 aldoxorubicin IV.
Period: Overall Study
Arm/Group | 250 mg/m^2 Aldoxorubicin | 350 mg/m^2 Aldoxorubicin
Started | 21 | 7
Completed (Completed defined as receiving at least one dose of study drug.) | 21 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 250 mg/m^2 Aldoxorubicin | 350 mg/m^2 Aldoxorubicin | Total
Number analyzed (Participants) | 21 | 7 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.29) | 54.2 (15.37) | 54.4 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 13 | 6 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 17 | 5 | 22
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 18 | 6 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete Response and Partial Response)
Description: ORR was defined as the proportion of patients with objective CR or PR by RANO working group criteria.
  CR: required all the following: complete disappearance of all enhancing measurable/ non-measurable disease sustained for at least 4 weeks; no new lesions; stable or improved non-enhancing (T2/FLAIR) lesions; patients must be off corticosteroids (or on physiologic replacement doses only); and stable or improved clinically. Patients with non-measurable disease only cannot have a CR.
  PR: Requires all of the following: ≥50% decrease compared with baseline sustained for at least 4 weeks; no PD of non-measurable disease; no new lesions; stable or improved non-enhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan; the corticosteroid dose at the time of the scan evaluation should be no greater than the dose at the time of the baseline scan; and stable or improved clinically. Patients with non-measurable disease only can't have a PR.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- 250 mg/m^2 Aldoxorubicin: Subjects received 250 mg/m^2 aldoxorubicin IV.
  250 mg/m^2 aldoxorubicin
- 350 mg/m^2 Aldoxorubicin: Subjects received 350 mg/m^2 aldoxorubicin IV.
  350 mg/m^2 aldoxorubicin
Arm/Group | 250 mg/m^2 Aldoxorubicin | 350 mg/m^2 Aldoxorubicin
Number analyzed (Participants) | 21 | 7
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: AEs that occurred during the clinical trial, starting at the time of the initial study drug infusion, and the follow-up period were recorded on the appropriate AE page of the CRF. All SAEs that occurred during the course of the study or within 30 days of the last administration of study medication were reported. The SAE reporting period ended if the subject began an alternative therapy within 30 days of the last administration of study drug. The expected duration is 24 months.
Arm/Group | 250 mg/m^2 Aldoxorubicin | 350 mg/m^2 Aldoxorubicin
All-Cause Mortality (participants affected / at risk) | 16/21 | 7/7
Serious Adverse Events (participants affected / at risk) | 6/21 | 2/7
Other Adverse Events (participants affected / at risk) | 21/21 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg/m^2 Aldoxorubicin (N=21) | 350 mg/m^2 Aldoxorubicin (N=7)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Cerebrolvascular accident (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg/m^2 Aldoxorubicin (N=21) | 350 mg/m^2 Aldoxorubicin (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Tachycardia (Cardiac disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Papilloedema (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Mouth ulcerations (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 5
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 2 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3
Catheter site pain (General disorders) | 5 | 0
Fatigue (General disorders) | 14 | 7
Infusion site reaction (General disorders) | 4 | 1
Mucosal inflammation (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Candida infection (Infections and infestations) | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 1
Oral candidiasis (Infections and infestations) | 3 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Hematocrit decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0
White blood cells count decreased (Investigations) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Aphasia (Nervous system disorders) | 2 | 1
Brain oedema (Nervous system disorders) | 2 | 1
Cognitive disorder (Nervous system disorders) | 2 | 0
Coordination abnormal (Nervous system disorders) | 1 | 1
Dysguesia (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 3
Hemiparesis (Nervous system disorders) | 5 | 1
Memory impairment (Nervous system disorders) | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 2
Somnolence (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 2
Visual field defect (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 3 | 0
Mood swings (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Allopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Nail bed disorder (Skin and subcutaneous tissue disorders) | 1 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT02014844/Prot_SAP_000.pdf